CLINICAL TRIAL: NCT05887245
Title: Znaczenie Kliniczne przywierającego tłuszczu okołonerkowego u pacjentów Poddawanych Resekcji Guza Nerki
Brief Title: Clinical Significance of Adherent Perinephric Fat in Patients Undergoing Partial Nephrectomy
Status: Active, not recruiting | Type: Observational
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor
Other Study IDs: nr 21/2023
Record Dates: First submitted 2023-05-18; First posted 2023-06-02 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-11

CONDITIONS: Renal Cell Carcinoma; Kidney Neoplasm; Urologic Neoplasms; Urogenital Neoplasms; Kidney Diseases
Keywords: Partial Nephrectomy; Adherent Perinephric Fat
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to gain a better understanding of the phenomenon of adherent perinephric fat (APF), which occurs in some patients undergoing partial nephrectomy (PN). This phenomenon, so-called "toxic fat", is a commonly recognized problem among urologists, but its significance has not yet been fully understood. The study aims to identify new clinical risk factors for APF occurrence and evaluate its impact on functional, perioperative, and oncological treatment outcomes. The study will be conducted on patients who are qualified for PN surgery. Prior to the surgical procedure, venous blood will be collected, which will be used for various measurements, such as blood morphology, kidney parameters, inflammation markers, liver function tests, glucose, and lipid profile. In addition, medical data will be collected concerning the patient's overall health, observed changes in the kidney, perioperative course, hospitalization, and histopathological characteristics of the tumor. After treatment, patients will be followed up for up to 60 months. The knowledge gained from this study can significantly assist in making decisions about surgical treatment and thus contribute to improving the treatment outcomes of patients with kidney tumors.

DETAILED DESCRIPTION:
Patients qualified for partial nephrectomy surgery based on radiological diagnosis of kidney tumor will be prospectively identified. Thirty milliliters of venous blood will be collected one day prior to the procedure. Blood samples will be sent to the laboratory, where, in addition to the standard preoperative tests (blood count, creatinine, urea, fasting glucose), the following parameters will be determined: C-reactive protein, ferritin, total cholesterol, low density lipoprotein, high density lipoprotein, and triglycerides. At the time of patient enrollment in the study, a clinical and demographic interview will be conducted. In addition, the hospital's electronic medical records will be used to obtain preoperative conventional imaging test results related to tumor characteristics. During the treatment, perioperative parameters will also be collected, including the presence of APF defined intraoperatively by the surgeon. APF is defined as "perinephric fat adherent to the renal parenchyma, making renal dissection difficult" with the presence defined by the surgeon as 1 - present, 0 - absent. The patient's participation in the study will not affect the type or technique of the surgery, and therefore, the risk of complications. After obtaining the histopathological result, data regarding the removed tumor will be collected. During the observation period (6, 12, 24, and 60 months after treatment), oncological and functional outcomes will be assessed and recorded. The observation will be conducted according to the treating physician's recommendations, in accordance with current medical knowledge, and its modification is not the subject of this study. Patient data will be collected and stored in an electronic database. The assessment of the relationship between the various blood parameters, demographic characteristics (age, gender), clinical characteristics (such as BMI, presence of metabolic syndrome, tumor size), and the presence of APF will be performed using univariate analysis (Chi-square, univariate logistic regression) and multivariate analysis (logistic regression models). When evaluating the impact of APF on perioperative and oncological outcomes, confounding variables (such as tumor stage, surgical method, surgeon) will be taken into account when creating predictive models.

ELIGIBILITY:
Inclusion Criteria:

* Patients qualified for partial nephrectomy by open, laparoscopic, or robotic method
* Tumor stage cT1a-cT1b according to Tumour Node Metastasis classification
* Age ≥ 18 years
* Written consent to participate in the study

Exclusion Criteria:

* Patient does not give consent to participate in the study
* Patients with recurrent kidney cancer, or who have undergone other surgeries within the kidney
* Lack of preoperative imaging available for assessment
* Missing medical documentation that prevents data analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a radiological diagnosis of kidney tumor referred for surgical treatment with partial nephrectomy will be eligible.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical risk factors for the occurrence of adherent perinephric fat in patients undergoing partial nephrectomy. | Data gathered in the pre-operative period. Blood samples collected one day prior to surgery.
  The following variables will be evaluated:
  1. Anthropometric (sex; age in years; weight in kilograms; height in centimeters; waist circumference in centimeters) and comorbidity data (assessed with Charlson Comorbidity Index, 0-24).
  2. Laboratory test results (C-reactive protein in mg/l; total cholesterol in mg/dl; triglycerides in mg/dl; high density lipoprotein in mg/dl; low density lipoprotein in mg/dl; ferritin in ng/ml; fasting glucose in mg/dl; creatinine in mg/dl; glomerular filtration rate calculated with the Modification of Diet in Renal Disease equation in ml/min/1,73 m²; white blood cell in G/l; lymphocyte in G/l; monocyte in G/l; hemoglobin in g/dl; platelets in G/l; neutrophil in G/l).
  3. Imaging data and tumor features (maximum tumor diameter in millimeters; perirenal fat thickness in millimeters; Mayo Adhesive Probability score, 0 - 5; RENAL Nephrometry Score, 4 - 12).

SECONDARY OUTCOMES:
Evaluation of the impact of adherent perinephric fat on functional, perioperative, and oncological treatment outcomes. | Data gathered in the post-operative period. Observation period 6,12, 24, and 60 months after treatment.
  The following variables will be evaluated:
  1. Peri-operative (operative time in minutes; warm ischemia time in minutes; estimated blood loss in minutes) and post-operative data (complications assessed with Clavien-Dindo Classification, I-V).
  2. Tumor histopathological characteristics (tumor type; maximum tumor diameter in millimeters; tumor stage according to the Tumour Node Metastasis classification; Fuhrman grade 1-4; surgical margins 0-1).
  3. Oncological (recurrence-free survival in months, overall survival in months), functional (estimated glomerular function change in ml/min/1,73 m²) outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sławomir Poletajew, Prof., Principal Investigator — Second Department of Urology, Centre of Postgraduate Medical Education
Locations (1):
- European Health Centre, Second Department of Urology, Centre of Postgraduate Medical Education, Otwock, Poland